CLINICAL TRIAL: NCT03562468
Title: A Randomized, Double-Blind, Crossover Study to Assess the Effects of Nicotinamide Riboside on Cognitive Function, Mood and Sleep in Older Adult Men and Women
Brief Title: A Study by ChromaDex to Assess the Effects of TRU NIAGEN on Cognitive Function, Mood and Sleep in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChromaDex, Inc. (Industry)
Collaborators: Midwest Center for Metabolic and Cardiovascular Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MB-1801
Record Dates: First submitted 2018-05-25; First posted 2018-06-19 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Cognitive Function; Mood; Sleep
Keywords: Nicotinamide riboside; NAD; TRU NIAGEN
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Treatments will be administered daily as 4 capsules in a double-blind, randomized, crossover manner for three 8-week treatment periods. Each subject will receive one placebo and two active treatments in a crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study site will be provided placebo and TRU NIAGEN capsules, each labeled with the protocol number, blinded product code, expiration date, batch number, the statement "For Investigational Use Only" and a space to write the subject's initials, screen and date dispensed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Each subject will be randomly assigned to receive placebo for an 8-week treatment period. Subjects will be instructed to take two capsules (placebo) in the morning with breakfast and two capsules (placebo) in the evening with dinner. At the end of each 8-week treatment period subjects will crossover to the next treatment group until all three treatment periods have been completed at 24 weeks.
  Interventions: Dietary Supplement: Placebo
- TRU NIAGEN (nicotinamide riboside) 300 mg/day (Experimental): Each subject will be randomly assigned to receive 300 mg/day of TRU NIAGEN (nicotinamide riboside) for an 8-week treatment period. Subjects will be instructed to take two capsules of TRU NIAGEN in the morning with breakfast and two capsules of TRU NIAGEN in the evening with dinner. At the end of each 8-week treatment period subjects will crossover to the next treatment group until all three treatment periods have been completed at 24 weeks.
  Interventions: Dietary Supplement: 300 mg/day of TRU NIAGEN (nicotinamide riboside)
- TRU NIAGEN (nicotinamide riboside) 1000 mg/day (Experimental): Each subject will be randomly assigned to receive 1000 mg/day of TRU NIAGEN (nicotinamide riboside) for an 8-week treatment period. Subjects will be instructed to take two capsules of TRU NIAGEN in the morning with breakfast and two capsules of TRU NIAGEN in the evening with dinner. At the end of each 8-week treatment period subjects will crossover to the next treatment group until all three treatment periods have been completed at 24 weeks.
  Interventions: Dietary Supplement: 1000 mg/day of TRU NIAGEN (nicotinamide riboside)

INTERVENTIONS:
Dietary Supplement: 300 mg/day of TRU NIAGEN (nicotinamide riboside) — Treatment with 300 mg/day of TRU NIAGEN (nicotinamide riboside) will be administered daily as 4 capsules in a double-blind, randomized, crossover manner for three 8-week treatment periods. Each subject will receive one placebo and two active treatments in a crossover design. The two active treatments are 300 mg/d TRU NIAGEN (nicotinamide riboside) and 1000 mg/d TRU NIAGEN (nicotinamide riboside).
  Other Names: Niagen, the active ingredient in TRU NIAGEN
  Arms: TRU NIAGEN (nicotinamide riboside) 300 mg/day
Dietary Supplement: 1000 mg/day of TRU NIAGEN (nicotinamide riboside) — Treatment 1000 mg/day of TRU NIAGEN (nicotinamide riboside) will be administered daily as 4 capsules in a double-blind, randomized, crossover manner for three 8-week treatment periods. Each subject will receive one placebo and two active treatments in a crossover design. The two active treatments are 300 mg/d TRU NIAGEN (nicotinamide riboside) and 1000 mg/d TRU NIAGEN (nicotinamide riboside).
  Other Names: Niagen, the active ingredient in TRU NIAGEN
  Arms: TRU NIAGEN (nicotinamide riboside) 1000 mg/day
Dietary Supplement: Placebo — Treatment with placebo capsules will be administered daily as 4 capsules in a double-blind, randomized, crossover manner for three 8-week treatment periods. Each subject will receive one placebo and two active treatments in a crossover design. The two active treatments are 300 mg/d TRU NIAGEN (nicotinamide riboside) and 1000 mg/d TRU NIAGEN (nicotinamide riboside).
  Arms: Placebo

SUMMARY:
The sponsor of this study is ChromaDex, Inc. This is a double-blind, randomized, crossover study to investigate the effects of 300 mg/d and 1000 mg/d TRU NIAGEN (nicotinamide riboside) compared to a placebo control on cognitive function, mood and sleep in men and women over 55 years of age. The trial is managed by Midwest Center for Metabolic and Cardiovascular Research.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, ≥55 years of age.
2. Subject has a BMI of 18.50 to 34.99 kg/m2.
3. Subject has a score of ≥80 on executive function at screening. One re-test will be allowed for subjects who require additional instruction on the CNS VS test battery.
4. Subject is willing to maintain usual diet and physical activity patterns.
5. Subject has no plans to change smoking habits during the study period.
6. Subject is willing to limit alcohol consumption to no more than one serving of alcohol per day (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor) and will abstain from consuming 2 h prior to retiring for the evening for the duration of the study.
7. Subject is willing to limit consumption of caffeine-containing beverages/foods/products to no more than 400 mg daily, with all caffeine consumption occurring prior to 6 pm.
8. Subject is willing to fast (8 - 15 h, target 10 h, water only) prior to each clinic visit.
9. Subject has no difficulties swallowing capsules.
10. Subject is willing and able to attend all clinic visits.
11. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator and is willing to complete study procedures.

Exclusion Criteria:

1. Individual has history or presence of a clinically significant (in the opinion of the Investigator) psychiatric disorder or neurologic disease including epilepsy, cerebrovascular disturbance or traumatic injury.
2. Individual has a history of diagnosed clinical depression in the prior 2 years, or a score ≥20 (defined as moderate-to-severe depression) on the Beck Depression Inventory-II administered at visit 1 (week -1).
3. Individual is currently diagnosed with dementia and/or has a score <24 on the Mini Mental State Questionnaire administered at visit 1 (week -1).
4. Uncorrected abnormal vision that in the opinion of the Investigator would impair the subject's ability to complete the computerized testing (including but not limited to nearsightedness, farsightedness, and color blindness).
5. Individual has a clinically important active endocrine, cardiovascular, renal, hepatic, pulmonary, pancreatic, neurologic or biliary disorder.
6. Individual has a history of a cardiovascular event or revascularization procedure within 6 months of visit 1 (week -1).
7. Individual has a diagnosis of type I diabetes mellitus. Type 2 diabetes mellitus is excluded if the individual has experienced initiation of or a dosage change in diabetes medication(s) within 2 months of visit 1 (week -1), or has significant co-morbidities as determined by the study physician.
8. Insulin for the treatment of Type I or Type 2 diabetes mellitus is exclusionary.
9. Individual has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg).
10. Individual has a recent history (prior 5 years) or the presence of cancer other than non-melanoma skin cancer.
11. Individual has a history or presence of a chronic pain condition requiring regular use of opioid therapy.
12. Individual has a recent history or strong potential for drug or alcohol abuse defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1 ½ oz distilled spirits).
13. Individual has a history of unconventional sleep patterns (e.g., night shift) or chronic insomnia (at least 3 d/week over the past month), a diagnosed sleep disorder, or a chronic medical condition with the potential to impact energy/fatigue levels.
14. Individuals taking any form of niacin >25 mg/d and any use of nicotinamide riboside within 2 weeks of visit 1 (week -1).
15. Individual is a heavy consumer of caffeinated beverages (>400 mg/d within 2 weeks of visit 1).
16. Individual has a history of using psychotropic medications (including antidepressants and tranquilizers), stimulant medications, and/or narcotics within 4 weeks of visit 1 (week -1).
17. Individual has used sleep aid medications, supplements, and/or products, including antihistamines, within 2 weeks of visit 1 (week -1) A washout prior to screening is allowed).
18. Individual has a known allergy to any ingredients in the study products.
19. Individual is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to use of a medically approved form of contraception throughout the study period.
20. Subject has an active infection or has used antibiotics within 5 d of any clinic visit. For those with an active infection and/or using antibiotics, subjects must wait at least 5 d after the infection resolves or antibiotic use is complete. The test period will be extended for completion in these cases.
21. Subject has been exposed to any non-registered drug product within 30 d of visit 1 (week -1).
22. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
The primary comparison will be the low dose (300 mg/d nicotinamide riboside) condition to the placebo condition for the change from baseline to the end of each relevant treatment period. | 8 weeks
  The primary outcome variable will be the difference between treatments in the change from baseline (defined as visit 2 value for each of the three treatment periods) in executive function measured with the CNS Vital Signs test battery, using the standard score.

CONTACTS AND LOCATIONS:
Locations (1):
- MB Clinical Research, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No